CLINICAL TRIAL: NCT00495378
Title: Retrospective Review of Alternate PROCRIT Dosing In Patients With Chemotherapy Related Anemia
Brief Title: RAPID-2. A Study to Evaluate the Effectiveness of Alternate Dosing of PROCRIT (Epoetin Alfa) in Maintaining Hemoglobin Levels in Patients With Chemotherapy Related Anemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was stopped due to slow enrollment after enrolling 25 of 200 patients.
Sponsor: Ortho Biotech Products, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005128
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2007-06

CONDITIONS: Chemotherapy; Cancer; Anemia
Keywords: PROCRIT; Epoetin alfa; chemotherapy related anemia
MeSH Terms: conditions — Neoplasms; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study was to determine if alternate dosing of Epoetin alfa was effective in maintaining hemoglobin levels in patients with chemotherapy related anemia.

DETAILED DESCRIPTION:
This was a retrospective chart review of patients with chemotherapy related anemia. Two hundred (200) patients with chemotherapy related anemia were to have received PROCRIT (Epoetin alfa) on a weekly schedule (e.g., once every week or more frequently) for at least 4 weeks, followed by a maintenance PROCRIT (Epoetin alfa) schedule of less frequent dosing (e.g. once every 2 weeks, once every 3 weeks, or once every 4 weeks) for at least 6 weeks. Hemoglobin response and maintenance of initial treatment phase hemoglobin with alternate doses of PROCRIT (Epoetin alfa) were to be evaluated.Study sites were to record data in a Case Report Form which would then be entered into a database. Data was to be recorded, starting with the PROCRIT (Epoetin alfa) initiation phase (at least 4 weeks duration), and extending through at least 6 weeks of maintenance therapy. A minimum of 20 study sites were to be enrolled in the data collection process.Data obtained was to be analyzed to reflect alternate dosing patterns of PROCRIT (Epoetin alfa) therapy. The frequency and percentage of patients receiving each dosing regimen were to be summarized. Hemoglobin response and maintenance of initial treatment phase hemoglobin with alternate doses of PROCRIT (Epoetin alfa) were to be evaluated. If PROCRIT (Epoetin alfa) was discontinued, the time and reason(s) for discontinuation were to be recorded.

Patients were to have received PROCRIT (Epoetin alfa) subcutaneous injection on a weekly schedule (e.g., once every week or more frequently) for at least 4 weeks, followed by a maintenance PROCRIT (Epoetin alfa) schedule of less frequent dosing (e.g. once every 2 weeks, 3 weeks, or 4 weeks) for at least 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chemotherapy related anemia
* Patients with a diagnosis of malignancy
* Patients with initial weekly PROCRIT (Epoetin alfa) therapy for at least 4 weeks
* Patients must have received PROCRIT (Epoetin alfa) maintenance therapy with less frequent dosing (e.g. every 2 weeks, every 3 weeks, every 4 weeks) for at least 6 weeks immediately following once weekly dosing.

Exclusion Criteria:

* No previous diagnosis of hemolytic anemia or myelodysplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-11; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Frequency and percentage of subjects in each dosing regimen will be summarized. Hemoglobin (Hb) response and maintenance of initial treatment phase Hb with alternate doses of Epoetin alfa. Time and reasons for discontinuing Epoetin alfa.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech, Inc.

REFERENCES:
- See also: For FDA Approved Product labeling, refer to the following link:http://www.accessdata.fda.gov/scripts/cder/drugsatfda/ — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/
- See also: Additional information is provided at the following link:http://dailymed.nlm.nih.gov/dailymed/about.cfm — http://dailymed.nlm.nih.gov/dailymed/about.cfm